CLINICAL TRIAL: NCT06051370
Title: Ultrasound-guided Glenohumeral Versus Subacromial Steroid Injections for Impingement Syndrome With Mild Stiffness: A Randomized Controlled Trial
Brief Title: Glenohumeral Versus Subacromial Steroid Injections for Impingement Syndrome With Mild Shoulder Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stiff Impinge - GH vs SA
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Impingement Syndrome; Adhesive Capsulitis of Shoulder
Keywords: Glenohumeral injection; Subacromial injection; Ultrasound-guided injection; Steroid injection
MeSH Terms: conditions — Shoulder Impingement Syndrome; Bursitis | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Study group underwent ultrasound-guided posterior approach of glenohumeral space injection for impingement syndrome with mild stiffness of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine, 7 mL normal saline.
  Control group underwent ultrasound-guided anterolateral approach of subacromial space injection for impingement syndrome with mild stiffness of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine, 7 mL normal saline.
Who Masked: Participant, Outcomes Assessor
Masking Description: A final number of 51 patients were enrolled in the trial and randomly assigned to either the glenohumeral ultrasound-guided injection group (Group GH) or the subacromial ultrasound-guided injection group (Group SA). Double-blinded randomization was performed by an independent nurse using a computer-generated random sequence. A musculoskeletal radiologist, blinded to group allocation, performed the diagnostic ultrasound and MRI interpretations. A blinded orthopaedic resident and nurse carried out the physical examination and clinical scoring.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glenohumeral injection (Experimental): Ultrasound-guided posterior approach of glenohumeral space injection for impingement syndrome with mild stiffness of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine, 7 mL normal saline.
  Interventions: Procedure: Ultrasound-guided glenohumeral space triamcinolone, lidocaine and saline injection
- Subacromial injection (Active Comparator): Ultrasound-guided anterolateral approach of subacromial space injection for impingement syndrome with mild stiffness of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine, 7 mL normal saline.
  Interventions: Procedure: Ultrasound-guided subacromial space triamcinolone, lidocaine and saline injection

INTERVENTIONS:
Procedure: Ultrasound-guided glenohumeral space triamcinolone, lidocaine and saline injection — Using a 21-gauge spinal needle, the predefined steroid solution was injected under ultrasound guidance using 5- to 13-MHz linear probe into the glenohumeral space through the posterior approach
  Arms: Glenohumeral injection
Procedure: Ultrasound-guided subacromial space triamcinolone, lidocaine and saline injection — Using a 21-gauge spinal needle, the predefined steroid solution was injected under ultrasound guidance using 5- to 13-MHz linear probe into the subacromial space through the anterolateral approach
  Arms: Subacromial injection

SUMMARY:
A prospective randomized controlled trial enrolled 51 patients diagnosed with shoulder impingement syndrome and mild stiffness.

Patients were randomly assigned to two groups: the glenohumeral injection group (Group GH) or the subacromial injection group (Group SA). After the final follow-up, 48 patients (24 in each group) were included for analysis Using ultrasound guidance, a solution containing 1mL of triamcinolone, 4mL of 1% lidocaine, and 7mL of 0.9% normal saline was injected into either the glenohumeral or the subacromial space. The following assessments were conducted at baseline and during follow-up visits at weeks 3, 7, and 13: ROM measurements for forward elevation, external rotation, and internal rotation; clinical scores including VAS, ASES, and Constant.

DETAILED DESCRIPTION:
Patient Enrollment Following approval from the Institutional Review Board and in compliance with the Declaration of Helsinki, a prospective randomized controlled trial was conducted from January 2013 to June 2014, involving 56 patients diagnosed with shoulder impingement syndrome with mild stiffness. Impingement syndrome was diagnosed based on positive Hawkin's sign and radiographic findings (rotator cuff with intact continuity but tendinosis confirmed by MRI or ultrasound, with a possible subacromial enthesophyte). "Mild" stiffness was defined in this study as a degree of stiffness that permits activities of daily activity but still often causes endpoint ROM pain. It was specified as meeting two or more of the following criteria in shoulder range of motion both passive and active: abduction between 110˚ and 150˚, forward elevation between 120˚ and 140˚, external rotation at the side between 30˚ and 50˚, and internal rotation at 90˚ of abduction between 30˚ and 50˚.

Patients were excluded from the study if they (1) refused to undergo ultrasound-guided injection, (2) were diagnosed with a rotator cuff tear, calcific tendinosis, or biceps pathology, (3) had a history of operation, fracture, or nerve injury of the shoulder, or (4) received treatment apart from the protocol during the study. A final number of 51 patients were enrolled in the trial and randomly assigned to either the glenohumeral ultrasound-guided injection group (Group GH) or the subacromial ultrasound-guided injection group (Group SA). Double-blinded randomization was performed by an independent nurse using a computer-generated random sequence. A musculoskeletal radiologist (M. S. H.) with over 20 years of experience performed the diagnostic ultrasound and MRI interpretations. A shoulder specialist (J.-T. H.) with more than 10 years of experience performed the ultrasound-guided injections. A blinded orthopaedic resident and nurse carried out the physical examination and clinical scoring. After the final follow-up, 48 patients (24 in each group) were eligible for analysis

Treatment and Follow-up Protocol Diagnostic ultrasound was first done using a 5- to 12-MHz linear probe (Philips Healthcare, Bothell, WA) to rule out shoulder pathology other than impingement syndrome. Using a 21-gauge spinal needle, a solution of 1mL triamcinolone, 4mL 1% lidocaine, and 7mL 0.9% normal saline was injected under ultrasound guidance using 5- to 13-MHz linear probe (GE Healthcare, Chicago, IL) into either the glenohumeral space through the posterior approach or the subacromial space through the anterolateral approach. Patients were then seen in 3, 7, and 13 weeks after the injection. Oral aceclofenac 100 mg twice daily and omeprazole 20mg once daily were prescribed during follow-up. Stretching exercises in all ranges of motions commenced in the third week. Using a wand, patients were instructed to passively stretch their shoulders to an endpoint where pain is felt and keep that position for at least 30 seconds, five sessions a day, five minutes per session. Rubber band strengthening was added in the seventh week, concentrating on external rotation at the side. Using a rubber band (Thera-band, Hygienic Corp., Akron, OH) tied into a loop, the patients were educated to keep maximum painless external rotation for 30 seconds, five sessions a day, five minutes per session. The tension of the rubber band was decided depending on the patients' ability to keep the painless maximum rotation for thirty seconds.

Clinical Assessment and Data Collection Patient information, including age, sex, duration of symptoms, affected side, and hand dominance, was recorded. The following assessments were performed at baseline and at follow-up visits in weeks 3, 7, and 13: range of motion (ROM) in forward elevation (FE), external rotation at the side (ER), and internal rotation at 90˚ of abduction (IR), pain visual analog scale (pVAS), American Shoulder and Elbow Surgeons (ASES) score, and the Constant-Murley (Constant) score. The ASES score was chosen as it was much verified to best reflect the activities of daily living, while strength was evaluated through the Constant score Improvement in ROM was calculated by subtracting the pre-injection measurements from the measurements at each follow-up visit.

Statistical Analysis A power analysis determined that a sample size of 42 patients (21 per group) would be sufficient to have an 80% statistical power to detect a significant difference in the improvement of the Constant score between pre-injection and 7-week post-injection, with a two-sided α level of 0.05. An effect size of 0.89 was assumed based on the mean difference and standard deviation of improvement in the Constant score between pre-injection and 7-week post-injection in a pilot study of 20 patients.

Normal distribution was checked using the Kolmogorov-Smirnov test. The independent-samples t test or the Mann-Whitney U test were used to analyze continuous data, while the paired-sample t test was used for intra-group comparison of serial measurements. Categorical data were analyzed using Pearson's chi-squared test. Continuous data were described as mean ± SD, and categorical data as a percentage. Analyses were performed using SPSS version 25 (IBM Corporation, Armonk, NY), and a P-value below 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with shoulder impingement syndrome with mild stiffness.
* Impingement syndrome diagnosed based
* Positive Hawkin's sign and
* Rotator cuff with intact continuity but tendinosis in MRI or US
* Possible subacromial enthesophyte
* Mild stiffness was defined as a degree of stiffness that permits activities of daily activity but still often causes endpoint ROM pain
* Meeting two or more of the following ROM both active & passive
* Abduction between 110˚ and 150˚
* Forward elevation between 120˚ and 140˚
* External rotation at the side between 30˚ and 50˚
* Internal rotation at 90˚ of abduction between 30˚ and 50˚.

Exclusion Criteria:

* Refused to undergo ultrasound-guided injection
* Diagnosed with a rotator cuff tear, calcific tendinosis, or biceps pathology
* History of operation, fracture, or nerve injury of the shoulder
* Received treatment apart from the protocol during the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-01-12 (Actual); Primary Completion 2014-03-17 (Actual); Study Completion 2014-06-18 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) for pain | Change from the baseline at 13 weeks
  Patient-reported 0-10 scale of pain, 0: no pain, 10: very severe pain
Range of motion (ROM) | Change from the baseline at 13 weeks
  ROM in degrees, forward elevation (0-150), external rotation (0-90), and internal rotation (0-90)
American Shoulder and Elbow Surgeons (ASES) shoulder score | Change from the baseline at 13 weeks
  Patient-reported shoulder satisfaction score, 0-100, higher scores mean a better outcome.
Constant score | Change from the baseline at 13 weeks
  Patient-reported and healthcare provider-assessed shoulder satisfaction score, 0-100, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrison AK, Flatow EL. Subacromial impingement syndrome. J Am Acad Orthop Surg. 2011 Nov;19(11):701-8. doi: 10.5435/00124635-201111000-00006. PMID 22052646
- [Background] Namdari S, Yagnik G, Ebaugh DD, Nagda S, Ramsey ML, Williams GR Jr, Mehta S. Defining functional shoulder range of motion for activities of daily living. J Shoulder Elbow Surg. 2012 Sep;21(9):1177-83. doi: 10.1016/j.jse.2011.07.032. Epub 2011 Nov 1. PMID 22047785
- [Background] Mathews PV, Glousman RE. Accuracy of subacromial injection: anterolateral versus posterior approach. J Shoulder Elbow Surg. 2005 Mar-Apr;14(2):145-8. doi: 10.1016/j.jse.2004.06.012. PMID 15789007
- [Background] Wright RW, Baumgarten KM. Shoulder outcomes measures. J Am Acad Orthop Surg. 2010 Jul;18(7):436-44. doi: 10.5435/00124635-201007000-00006. PMID 20595136
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738